CLINICAL TRIAL: NCT02376933
Title: Phase 2 Study of Vertebral Augmentation and Radiotherapy in Painful or at Risk of Collapse Spinal Metastatic Cancer/Multiple Myeloma
Brief Title: Vertebral Augmentation and Radiotherapy of Collapse Spinal Metastatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the department; protocol transfer did not take place.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1300000562
Record Dates: First submitted 2015-02-20; First posted 2015-03-03 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Metastatic Cancers; Multiple Myeloma; Vertebral Fracture
Keywords: vertebral bodies; vertebral fracture; vertebral augmentation; radiotherapy; vertebroplasty; kyphoplasty
MeSH Terms: conditions — Neoplasms; Multiple Myeloma; Spinal Fractures | interventions — Vertebroplasty; Kyphoplasty; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vertebroplasty with Radiotherapy (Experimental): Vertebroplasty with Radiotherapy is given in either order. Radiotherapy dosage is at the discretion of the treating physician. Vertebroplasty is applied to fractured vertebrae.
  Interventions: Procedure: Vertebroplasty; Radiation: Radiotherapy

INTERVENTIONS:
Procedure: Vertebroplasty — Under imaging guidance, a fractured vertebral body is stabilized with injected bone cement.
  Other Names: kyphoplasty
Radiation: Radiotherapy — Radiotherapy of metastatic lesions to the spine.

SUMMARY:
Vertebral augmentation with radiotherapy to increase the functional status and quality of life for patients with vertebral body metastatic cancers.

DETAILED DESCRIPTION:
The study quantifies the reduction of pain and changes in quality of life associated with vertebral augmentation. This study is conducted in patients with metastatic cancer or multiple myeloma involving the spine. This study addresses the value of vertebral augmentation in combination with radiotherapy in the setting of cancer to the spine. The patient's pain, overall quality of life, and fracture development/avoidance will be compared to patients treated only with radiotherapy in the past.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic disease to the vertebra or multiple myeloma
* Negative pregnancy test within 2 weeks prior to registration
* Life expectancy of >= 3 months and Karnofsky performance status (KPS) score >= 40
* Pain scale score >=5
* Pain at involved vertebral body not adequately controlled
* Osteolysis of vertebral bodies
* Must agree to practice adequate means of birth control
* Must sign informed consent prior to study entry
* Must be able to understand the English language
* Absence of any serious cognitive or psychiatric problems potentially hampering compliance with the study and follow-up schedule.

Exclusion Criteria:

* Spinal Cord Compression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2016-08-10 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krisha Howell, MD, Principal Investigator — University of Arizona Radiation Oncology
Locations (1):
- University of Arizona, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vertebroplasty With Radiotherapy
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vertebroplasty With Radiotherapy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment From the Worst Pain Score on Brief Pain Inventory as Compared to Historical Radiation Therapy Oncology Group (RTOG) 9714 Study.
Description: Assessment of the patient's pain, activities and quality of life will be gathered from the patient in returning for follow-up or by contacting the patient by phone approximately 1 week following the completion of their first procedure, whether it be the vertebral augmentation or the radiotherapy (5 - 10 days following). Mandatory assessments include:
  - Worst Pain Score - Brief Pain Inventory (BPI) - The Worst Pain Assessment on the Brief Inventory Scale is an assessment tool of current pain intensity and pain intensity within the last 24 hours when not on pain control medications. 0 being no pain and 10 is the worst pain possible. See protocol attachments
Time Frame: 14 weeks
Population: Study terminated when PI left institution; data not collected.
Arm/Group | Vertebroplasty With Radiotherapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Activity Level Assessment From the Roland Morris Questionnaire (RDQ) and Karnofsky Performance Status (KPS)
Description: Roland-Morris Disability Questionnaire - The score of the RDQ is the total number of items checked - i.e. from a minimum of 0 (best) to a maximum of 24 (worst).
  Karnofsky Performance Status (KPS) - scale from 10 (moribund, fatal processes progressing rapidly) to 100 (normal, no complaints, no evidence of disease).
Time Frame: 14 weeks
Population: Study terminated when PI left institution; data not collected.
Arm/Group | Vertebroplasty With Radiotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Quality of Life Assessment From the EORTC QLQ C30 Questionnaire.
Description: EORTC QLQ-C30 (version 3) - The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning,a high score for the global health status / QoL represents a high QoL,but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Time Frame: 14 weeks
Population: Study terminated when PI left institution; data not collected.
Arm/Group | Vertebroplasty With Radiotherapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Fracture Rates Detected From X-rays.
Time Frame: 14 weeks
Population: Study terminated when PI left institution; data not collected.
Arm/Group | Vertebroplasty With Radiotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Vertebroplasty With Radiotherapy
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vertebroplasty With Radiotherapy (N=10)
Gastrointestinal - other (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vertebroplasty With Radiotherapy (N=10)
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 2
Flu-like syndrome (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT02376933/Prot_000.pdf